CLINICAL TRIAL: NCT02153138
Title: The Effect of Plant-based Diets (Vegetarian and Vegan) on Endothelial Function and Atherogenic Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TASMC-14-VN-0085-CTIL
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Other Endothelial Dystrophy
Keywords: vegetarian diet; vegan; cardiovascular diseases; endothelial function; carotid intima-media thickness
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endo-pat 2000 — The endo peripheral arterial tonometry (PAT) provides an index of endothelial function in two forms:
  1. The reactive hyperemia index (RHI) is the post-to-preocclusion PAT signal ratio in the occluded side, normalized to the control side and further corrected for baseline vascular tone.
  2. The logarithm RHI (LnRHI) is s similar index as RHI after natural log transformation with a matched cutoff. LnRHI provides better double-sided distribution than RHI and one that is closer to normal distribution
Device: carotid intima media thickness Ultrasound — cIMT is the distance between the intimal-luminal interface and the medial-adventitial interface. It will be studied by B-mode ultrasonography of the extracranial carotid arteries. A duplex system with a 7-10 megahertz (MHz) linear array multi-frequency transducer will be used.
Device: Dexa- Bone densitometer & Bone ultrasonometer System — A means of measuring bone mineral density and body composition by a dual energy X-ray absorptiometry (DEXA) machine

SUMMARY:
The investigators' hypothesis is that a plant-based diet may be beneficial if nutritional deficiencies will be corrected. The aims of the present proposal are to 1) study endothelial functions of subjects on well-defined vegetarian/vegan diets compared to age and sex matched omnivores (controls), and 2) study the differences in energy expenditure, body composition, overnight substrate utilization, blood work results, and levels of intracellular reactive oxygen species (ROS) and of adhesion molecules on the different diets.

DETAILED DESCRIPTION:
The serious doubts about the nutritional adequacy of vegetarian diets in the past were essentially put to rest by recent studies that suggested that plant-based diets are healthy and associated with lower risk of several chronic diseases. Nevertheless, various nutritional deficiencies have been identified, and it has been shown that individuals who follow different types of vegetarian/vegan diets may not experience the same effects on their health.

Working Hypothesis

1. Vegetarian/vegan diets will promote protection against cardiovascular risk factors if supplemented with possibly deficient nutrients.
2. There will a further protective effect and a greater number of differences between subjects following a vegetarian diet compared to those following a vegan diet.
3. Higher energy expenditure and lower and different caloric intake will promote a favorable difference in body composition (lower body fat) via a different substrate utilization expressed in the measured respiratory quotient (RQ).
4. Extra- and intracellular free radicals will be higher in subjects who adhere to vegetarian/vegan diets compared to omnivores.

Aims of the study

1. To study the effect of vegetarian/vegan diets on endothelial functions after correcting for modifying factors.
2. To study the effect of the above-mentioned plant-based diets on carotid intima-media thickness.
3. To study the differences in body composition, resting energy expenditure and over-night substrate utilization between the different diets.
4. To study the intracellular ROS of subjects following different diets.

ELIGIBILITY:
Inclusion Criteria:

* over 5 years' adherence to any type of diet
* age range 35-50 years
* BMI ≤32

Exclusion Criteria:

* smoking
* type I and II diabetes
* liver and kidney impairments
* cardiovascular diseases
* patients with tumors
* patients on medications which may affect cardiovascular parameters (including 5 phosphodiesterase inhibitors, beta blockers, ACE inhibitors and others)
* BMI >32 kg/m2.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
carotid intima-media thickness (cIMT) | 1 year
  measure the differences in the thickness of the carotid between the different diet group

SECONDARY OUTCOMES:
body composition | 1-year
  Measure the differences in body composition ( fat %, lean body mass) between the different diet groups

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center